CLINICAL TRIAL: NCT06455891
Title: MYCobiome Analysis in Atopic Dermatitis With Head and Neck Involvement
Acronym: MYCAH
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: SGZ-2020-13289; 2024-A00281-46 (Other: IDRCB ANSM)
Record Dates: First submitted 2024-05-07; First posted 2024-06-12 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Atopic Dermatitis
Keywords: Head and neck atopic dermatitis (HNAD); skin mycobiome; Immunity modulation
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Patients with generalized AD defined by AD skin lesion involved more or equal 50% of total body surface area with head and neck involvement. (15 patients)
- Group 2: Patients with head and neck AD (HNAD) defined by AD involving at least 80% of the head and neck area with or without AD involvement outside the head and neck area but <20% of total body surface area. (15 patients)
- Group 3: Healthy control without chronic skin disease. Healthy control will be recruited from non-atopic patients explored in ours departments for drug allergy after resolution of acute events. (15 healthy controls)

SUMMARY:
It is an open study, explorative, proof of concept study concerning mycobiota dysbiosis implication in AD patients with head and neck involvement.

DETAILED DESCRIPTION:
The aim of this study is to carry out an analysis of the mycobiome in the head and neck regions of 30 adults with Atopic dermatitis compared with 15 healthy controls.

patients and participants will be recruited from 2 centers Hôpital Tenon AP-HP (Pr A Soria) and CHU Lille (Pr D Staumont-Sallé) over a 12-month period.

Patient will be classified in 2 subgroups according to topography and body surface area involved by AD;

* Group 1: Generalized AD defined by AD skin lesion involved more or equal 50% of total body surface area with head and neck involvement. (15 patients)
* Group 2: Head and neck AD (HNAD) defined by AD involving at least 80% of the head and neck area with or without AD involvement outside the head and neck area but <20% of total body surface area. (15 patients) Group 3: Healthy control without chronic skin disease. Healthy control will be recruited from non-atopic patients explored in ours departments for drug allergy after resolution of acute events. (15 healthy controls) In the framework of consultation, medical examination with clinical assessment, non-invasive skin microbiota samples (3x2 skin ESwab) will be performed and a supplemental blood sample was collected (35 mL) for study of innate and adaptive immune response (see Diagram of the study summarising the chronology of the study). For each patient the end of participation in the study is achieved after the completion of swab and blood samples. No follow up is planned. Patients' participation is 1 day at maximum.

Skin samples will be used for study of Mycobiome by culture and MALDI-TOF and NGS analysis and Blood sample will be used for study of the immune innate and adaptative response.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years;
* Male or female;
* The diagnosis of atopic dermatitis (AD) is defined according to the criteria of UK Working Party with at least 3 of the following 5 criteria are present; history of flexural involvement, history of a dry skin, onset under the age of 2, personal history of asthma or allergic rhinitis, history of a pruritic skin condition, and visible flexural dermatitis.
* Generalized AD defined by AD involved ≥50% of total body surface area with head and neck involvement. Or HNAD defined by AD involving at least 80% of the head and neck area with or without AD involvement outside the head and neck area but <20% of total body surface area.
* With topical anti-inflammatory treatments for AD (including; topical steroids and/or topical tacrolimus)
* Free, informed and written consent, signed by the patient and the investigator before any examination required by the trial;
* Affiliation to social security scheme (beneficiary or assignee)
* Healthy control are the same age and sex.

Exclusion Criteria:

* Systemic or local antifungal therapy within 2 months before entry and during the study
* Systemic treatments for AD; including: ciclosporine, dupilumab and others AD biologics, methotrexate, JAK-inhibitors
* Generalized AD without head and neck involvement
* AD involved less than 50% of total body surface
* Head and neck AD with less than 80% of the head and neck area involved
* Head and neck AD with more than 20% of AD involvement outside the head and neck area
* Current participation in another biomedical research
* Patient with a measure of legal protection
* Psychiatric illness or any other concomitant chronic illness or addiction that could be interfere with the ability to meet the requirements of the protocol or provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult, age between 18 and 65 years with generalized and head and neck AD treated with topical steroids and/or topical tacrolimus for AD.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-06-16 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Description and comparison of head and neck mycobiome in AD patients, with generalized AD and HNAD, compared to head and neck mycobiome in controls. | 18 months
  To conduct a mycobiome analysis in the Head and Neck areas in adults with AD compared to healthy control using matrix-assisted laser desorption ionization time of ﬂight mass spectrometry (MALDI-TOF) after culture. An additional analysis of the mycobiome by next generation sequencing (NGS) will also be carried out.

SECONDARY OUTCOMES:
Lectins and gene polymorphism implicated in innate response to mycobiome in AD patients with head and neck involvement. 15 mL of blood will be collected. | 18 months
  Study the interaction between mycobiome dysbiosis and immune responses in AD patients with head and neck involvement 1.
Antifungal systemic immune response. | 18 months
  20 mL of blood will be collected for specific Ig A, G, M and E detection and analysis of adaptive immune response against the predominant fungi identified in mycobiome of AD patients with head and neck involvement in order to study the interaction between mycobiome dysbiosis and immune responses in AD patients with head and neck involvement 2

CONTACTS AND LOCATIONS:
Overall Officials: Angèle SORIA, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Tenon Hospital APHP dermatology and allergology department, Paris, France

REFERENCES:
- [Background] Morgan XC, Huttenhower C. Chapter 12: Human microbiome analysis. PLoS Comput Biol. 2012;8(12):e1002808. doi: 10.1371/journal.pcbi.1002808. Epub 2012 Dec 27. PMID 23300406
- See also: Bibliographic reference — https://CRAN.R-project.org/package=vegan